CLINICAL TRIAL: NCT00003225
Title: Phase I/II Trial to Evaluate Ethyol as a Protective Agent for Irinotecan (CPT-11) Toxicities in Patients With Advanced Colorectal Cancer
Brief Title: Amifostine Plus Irinotecan in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: ALZA (Industry)
Responsible Party: Diane Prager, MD / Principal Investigator, UCLA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066087; UCLA-HSPC-970304601B; ALZA-UCLA-HSPC-970304601B; NCI-G98-1390
Record Dates: First submitted 1999-11-01; First posted 2004-07-21 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Amifostine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ethyol plus Irinotecan (Experimental): Ethyol 740 mg/m2 will be administered intravenously over 10 minutes. 10 minutes after completion of the Ethyol infusion, Irinotecan 250 mg/m2 will be given over 90 minutes IV.
  Interventions: Drug: amifostine trihydrate; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: amifostine trihydrate — Ethyol 740 mg/m2 will be administered intravenously over 10 minutes. Administered every two weeks for 3 cycles.
  Other Names: Ethyol
Drug: irinotecan hydrochloride — 10 minutes after completion of the Ethyol infusion, Irinotecan 250 mg/m2 will be given over 90 minutes IV.
  Administered every 14 days for 3 cycles

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of amifostine plus irinotecan in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity profile of irinotecan and amifostine when administered together in patients with metastatic colorectal cancer. II. Assess the total dose of irinotecan received per 6 week course in these patients. III. Determine the incidence of irinotecan-induced leukopenia, neutropenia, and diarrhea in these patients. V. Determine the response rate for this patient population.

OUTLINE: This is an open label study. Amifostine is administered by 10 minute IV infusions. Irinotecan is administered by IV infusions 15 minutes after completion of amifostine. Treatment is repeated every 2 weeks for 6 weeks. This 6 week course is repeated in the absence of disease progression. Treatment may be delayed up to 2 weeks after a course to allow for recovery from toxic effects. Patients are followed at the end of study and at 30 days after study.

PROJECTED ACCRUAL: There will be 25-30 patients accrued into this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ECOG 0-2
* Life expectancy of at least 12 weeks
* Pathologically confirmed diagnosis of metastatic colorectal cancer
* Measureable disease
* Have not received therapy for cancer within 4 weeks of enrollment on study
* Prior radiation therapy to the pelvis for treatment of colorectal cancer is allowed. Radiation therapy delivered elsewhere is allowed as long as the patient has been off treatment for at least six weeks and measurable lesions are present outside the radiation field
* Pretreatment granulocyte count of > 1500/mm3, hemoglobin > 9.0 g/dL (without transfusion), and platelet count of > 100,000/um
* Serum creatinine < 2.0 mg/dL
* Adequate hepatic function as documented by a serum bilirubin < 2.0 mg/dL regardless of whether patients have liver involvement secondary to tumor. AST must be < 3x the upper limit of normal unless the liver is involved with tumor, in which case the AST must be < 5x institutional upper limit of normal

Exclusion Criteria:

* Prior therapy with Irinotecan
* Patients with any active or uncontrolled infection
* Patients with psychiatric disorders that would interfere with consent or follow-up
* Patients with a history of myocardial infarction within the previous six months, congestive heart failure, or cerebrovascular disease
* History of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis
* Patients with uncontrolled diabetes mellitus
* Any other sever concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Patients unable to stop taking antihypertensive medication 24 hour prior to administration of Ethyol (off x 1 day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1997-07; Primary Completion 2000-03 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity profile of Irinotecan and Ethyol when administered together on this schedule. | 12 weeks

SECONDARY OUTCOMES:
To assess the total dose of Irinotecan received per 6 week cycle | 6 weeks
To determine incidence of Irinotecan-induced leukopenia and neutropenia | 12 weeks
To determine the incidence of Irinotecan-induced diarrhea | 12 weeks
To determine the response rate for patients with metastatic colorectal carcinoma receiving Irinotecan and Ethyol on this dosing schedule (as measured by time response, duration of response time to progression, time of treatment failure survival). | 12 weeks
To determine the clinical benefit of intravenous Irinotecan and Ethyol in patients with colorectal cancer, as measured by performance status, analgesic consumption, quality of life and survival. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane Prager, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Wilshire Oncology Medical Group, Inc., Rancho Cucamonga, California